CLINICAL TRIAL: NCT05951907
Title: The Anesthetic Efficacy of Articaine as Buccal Injection Compared to Lidocaine Baccual and Palatal Injection for Maxillary Premolar Teeth Extraction A Randomized, Single-Blinded, Clinical Trial.
Brief Title: The Anesthetic Efficacy of Lidocaine and Articaine as Buccal Injection for Maxillary Premolar Teeth Extraction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Almustafa Qays Abdulkareem, ALMUSTAFA QAYS ABDULKAREEM, POST GRADUATE STUDENT,UNIVERSITY F BAGHDAD, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Extraction By Articaine
Record Dates: First submitted 2023-07-03; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Case-Control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): A control group in which the extraction of the maxillary premolar's teeth was carried out under buccal and palatal infiltration anesthesia with 1.8 mL 2% lidocaine hydrochloride with 1:80,000 epinephrine.
  Interventions: Procedure: Maxillary extraction with buccal and palatal injection
- study group (Experimental): A study group in which the extraction of the maxillary premolar's teeth proceeded under buccal without palatal infiltration anesthesia with 1.8 mL, 4% articaine hydrochloride with 1:100,000 epinephrine.
  Interventions: Procedure: Maxillary extraction without palatal injection

INTERVENTIONS:
Procedure: Maxillary extraction without palatal injection — Extraction of maxillary premolars by only buccal injection without palatal by using articaine 4% HCL with epinephrine (1:100,000)
  Arms: study group
Procedure: Maxillary extraction with buccal and palatal injection — Extraction of maxillary premolars by only buccal and palatal injection by using lidocaine 2 % HCL with epinephrine (1:80,000)
  Arms: control group

SUMMARY:
This study Is designed as a prospective randomized, single-blinded clinical trial. To evaluate The anesthetic efficacy of articaine as a buccal Injection for maxillary premolar teeth extraction, compared to lidocaine as a buccal and palatal injection.

DETAILED DESCRIPTION:
In the current study, the sample size (200) patients were distributed into two groups, group (A), 100 patients extracted upper premolar teeth by using 1.8 mL cartridges of 4% articaine hydrochloride with 1:100,000 epinephrine (Artheek, Colombia) as a buccal injection without palatal injection, and Group (B), 100 patients were removed upper premolar teeth by using Injectable local anesthetic agents included; 1.8 mL cartridges of 2% lidocaine hydrochloride with 1:80,000 epinephrine (Huons, Korea) as a buccal and palatal injection, the pain assessment after extraction was assessed by using (vas) visual analog scale, comparison between the outcomes by the two groups were evaluated, according to many variables (age, gender, extracted tooth, type of anesthesia, extraction duration).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 16 years old, including both genders.
2. Patients indicated for extraction of one of the maxillary premolar's teeth.

Exclusion Criteria:

1. Patients who were allergic to the local anesthetic agents used in this study.
2. Patients who presented with acute periapical infections.
3. Patients who required surgical extraction that entails flap reflection and bone removal.
4. Pregnant patients.
5. Patients with uncontrolled systemic diseases.
6. Patients are taking medications affecting pain assessment, like opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Pain during Extraction | Assessment of pain in the period during which the extraction has been made and up to 5 minutes after extraction of the tooth.
  In the current study the pain during extraction was assessed by using the Visual Analogue Scale (VAS 0-10 cm ) one of the most commonly used self-reporting measures of pain, it measures a characteristic that is believed to range across a continuum of values range from (0 no pain) to the end (10 un bearable pain) which is not easy to measure directly .

CONTACTS AND LOCATIONS:
Overall Officials: Hasanain A. Al-Jumaily, C.A.B.M.S, Study Director — College of Dentistry - University of Baghdad
Locations (1):
- Almustafa Qays, Baghdad, Almansour, Iraq